CLINICAL TRIAL: NCT06293989
Title: Efficacy and Safety of Intravenous Diazepam Given at 2 Different Doses Compared to Placebo in Acute Peripheral Vertigo: A Randomized Controlled Double Blinded Study
Brief Title: Efficacy and Safety of Intravenous Diazepam Given at 2 Different Doses Compared to Placebo in Acute Peripheral Vertigo
Acronym: Vertigo
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, PROFESSOR, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Emergency department
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Vertigo, Peripheral
Keywords: vertigo; diazepam; placebo
MeSH Terms: conditions — Vertigo | interventions — Diazepam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- diazepam 5 mg (Experimental): Medications will be diluted with 5 mL of normal saline solution slowly intravenously injected (over 5 minutes). The associate clinical research coordinator was responsible for preparation and dispensing the study drug.
  Interventions: Drug: Diazepam 5mg
- diazepam 10 mg (Experimental): Medications will be diluted with 5 mL of normal saline solution slowly intravenously injected (over 5 minutes). The associate clinical research coordinator was responsible for preparation and dispensing the study drug.
  Interventions: Drug: Diazepam 10 mg
- placebo (Experimental): Medications will be diluted with 5 mL of normal saline solution slowly intravenously injected (over 5 minutes). The associate clinical research coordinator was responsible for preparation and dispensing the study drug.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diazepam 5mg — For the intervention, patients will be randomly allocated into three groups. Each patient will be randomized to one of three treatment groups: diazepam 5 mg (5 mg/1 mL), . Medications will be diluted with 5 mL of normal saline solution slowly intravenously injected (over 5 minutes). The associate clinical research coordinator was responsible for preparation and dispensing the study drug. The investigators, treating physicians, nurses, and patients were blinded to the treatment.
  Other Names: diazepam(B)
  Arms: diazepam 5 mg
Drug: Diazepam 10 mg — For the intervention, patients will be randomly allocated into three groups. Each patient will be randomized to one of three treatment groups: diazepam10 mg (5 mg/1 mL), . Medications will be diluted with 5 mL of normal saline solution slowly intravenously injected (over 5 minutes). The associate clinical research coordinator was responsible for preparation and dispensing the study drug. The investigators, treating physicians, nurses, and patients were blinded to the treatment.
  Other Names: diazepam(C)
  Arms: diazepam 10 mg
Drug: Placebo — For the intervention, patients will be randomly allocated into three groups. Each patient will be randomized to one of three treatment groups:Placebo . Medications will be diluted with 5 mL of normal saline solution slowly intravenously injected (over 5 minutes). The associate clinical research coordinator was responsible for preparation and dispensing the study drug. The investigators, treating physicians, nurses, and patients were blinded to the treatment.
  Other Names: A
  Arms: placebo

SUMMARY:
This is prospective, randomised double-blind study that will be conducted in the emergency department of 3 university hospitals (FB Monastir, Sahloul Sousse, and FH Sousse) to compare the efficacy of two doses of diazepam (Valium®) and placebo for the relief of acute periphery vertigo in the ED

DETAILED DESCRIPTION:
This is prospective, randomised double-blind study that will be conducted in the emergency department of 3 university hospitals (FB Monastir, Sahloul Sousse, and FH Sousse) to compare the efficacy of two doses of diazepam (Valium®) and placebo for the relief of acute periphery vertigo in the ED. The study should be reviewed and receive approval from the institutional review board. Principles of the Helsinki Declaration are considered All patients should provide their informed consent prior to enrollment.

ELIGIBILITY:
Inclusion Criteria;

* patients between 18 and 70 years of age
* a chief complaint of acute peripheral vertigo (APV) (sensation of spinning, which was worsened by movement and sudden in onset) were eligible if the treating emergency physician diagnosed an episode of vertigo that was peripheral in nature.

Exclusion Criteria: -Patients aged > 70 years as central vertigo , -patients with a focal neurologic deficit, pregnancy, history of allergic reaction or contraindication to any of the test drugs, history of enrolment in a previous clinical drug trial,

* history of recent ingestion (within 24 hours) of a sedative, antihistamine, antipsychotic, or opioid,
* history of syncope or cardiac event, considerations of a central origin for vertigo -evidence of drug-induced vertigo or orthostatic hypotension -history of mental or neurological illness.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale (VAS)-3H | 3 hours
  the frequency of vertigo resolution defined as a reduction of at least 50% in VAS at 3-hour(VAS-3H) compared to baseline VAS (VAS baseline) during movement (VAS ambulation).

SECONDARY OUTCOMES:
the Delta-VAS | 3 hous
  the delta VAS was calculated as [(VAS baseline- VAS3H)/VAS baseline]*100
the time required to reach the resolution of the vertigo crisis | 3 hours
  the time required to reach the resolution of the vertigo crisis
Patients satisfaction | 3 hours
  patient satisfaction with likert scale
number of patients with adverse effects | 3 hours
  number of patients with adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Nouira semir, Pr, Study Director — University of Monastir